CLINICAL TRIAL: NCT05760001
Title: A Randomized Controlled Trial of Concentrated Investment in Black Neighborhoods to Address Structural Racism as a Fundamental Cause of Poor Child Health
Brief Title: The IGNITE for Kids Study on Concentrated Investment in Black Neighborhoods and Child Health and Well-Being
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 850178b
Record Dates: First submitted 2023-02-23; First posted 2023-03-08 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Financial Stress; Economic Problems; Environmental Exposure; Health Behavior; Health, Subjective; Mental Health Wellness
MeSH Terms: conditions — Financial Stress; Health Behavior

STUDY DESIGN:
Masking Description: The investigators are not masked. Our recruitment team will be masked until cluster recruitment is complete. The outcomes assessor will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): At the individual level, participants in the intervention arm will receive place-based and financial well-being interventions.
  These will include, at the individual level:
  * Tax preparation
  * Access to public benefits
  * Financial counseling and microgrants
  At the neighborhood level:
  * Abandoned house remediation
  * Trash cleanup
  * Vacant lot greening
  * Tree planting
  Interventions: Other: Assigned Interventions
- Control Arm (No Intervention): Participants in the control arm will not receive any of the listed interventions

INTERVENTIONS:
Other: Assigned Interventions — Financial well-being interventions:
  • Tax preparation; access to public benefits; financial counseling and microgrants
  Place-based interventions:
  • Vacant lot greening; abandoned house remediation; trash cleanup; tree planting
  Arms: Intervention Arm

SUMMARY:
Black children and adults in the United States fare worse across nearly every health indicator compared to White individuals. In Philadelphia, the location of this study, these health disparities result in a stark longevity gap, with average life expectancies in poor, predominantly Black neighborhoods being 20 years lower than in nearby affluent, predominantly White neighborhoods. The investigators will conduct a cluster randomized controlled trial (RCT) of a suite of place- based and financial-wellbeing interventions at the community, organization, and individual/household levels that address the social determinants of racial health disparities. At the community level, the investigators address underinvestment in Black neighborhoods by implementing vacant lot greening, abandoned house remediation, tree planting, and trash cleanup. At the organization level, the investigators partner with community-based financial empowerment providers to develop cross-organizational infrastructure to increase reach and maximize efficiency. At the individual/household levels, the investigators increase access to public benefits, financial counseling and tax preparation services, and emergency cash assistance. The investigators will test this "big push" intervention in 60 Black neighborhood micro-clusters, with a total of 480 children. The investigators hypothesize that this "big push" intervention will have significant impact on children's health and wellbeing.

DETAILED DESCRIPTION:
Black individuals in the United States fare worse than White individuals across almost every social, economic, and health indicator. The Black health disadvantage starts at birth, reflecting the cumulative toll of racialized social stressors and healthcare discrimination on maternal health and resulting in higher rates of pre-term birth and low birth weight. Black youth are disproportionately exposed to environmental toxins such as lead and adverse childhood events such as financial hardship and neighborhood violence. Black children also have higher rates of chronic disease, including asthma and diabetes. These and other forces result in inequities in child health and well-being and can also impact children's educational and earning potential. Furthermore, these inequities culminate in a stark racial longevity gap: in Philadelphia, the location of this study, life expectancy for people living in a poor, predominantly Black neighborhood is 20 years lower than for people living in a nearby affluent, predominantly White neighborhood.

The fundamental cause of these striking and pervasive disparities is structural racism - the confluence of deep historical, institutional, cultural, and ideological forces that unequally distribute resources and risks across racialized groups. Structural racism patterns health by affecting a range of interconnected, mutually reinforcing social determinants of health at the national, neighborhood, household, and individual levels. Most notably, longstanding, systematic disinvestment has resulted in highly segregated Black neighborhoods with dilapidated environmental conditions and severe economic insecurity within Black households, leading to a "feedback loop of concentrated racial disadvantage," all of which have been strongly tied to poor health.

Most interventions seeking to address racial health disparities focus on individual-level behaviors and outcomes, or individual channels by which structural racism harms health. However, by failing to address upstream social determinants, these interventions have had limited population level impact. A multi-level, multi-component intervention package focused on a range of social determinants of health is necessary to meaningfully address structural racism as a fundamental cause of racial health disparities. In this trial, we aim to implement such a multi-level, multi-component intervention and then evaluate its impact on child health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Child is between the ages of 3 and 17 years at the start of the trial (between the ages of 5 and 19 years at the end of the trial)
* Parent/caregiver is at least 18 years of age
* Parent/caregiver has the ability to communicate via text messaging
* Parent/caregiver is comfortable communicating in English
* Child is a permanent resident of the home where they are to be enrolled
* Parent/caregiver has knowledge of their household finances

Exclusion Criteria:

* Children who plan to move out of the study microcluster within 6 months
* Children whose caregivers are unable to fully consent and participate based on CC team assessment

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 221 (Actual)
Dates: Start 2023-06-10 (Actual); Primary Completion 2026-02-17 (Estimated); Study Completion 2026-02-17 (Estimated)

PRIMARY OUTCOMES:
Child Health Questionnaire Parent Form 28 (CHQ-PF28) Composite Score | 24 months
  Composite index using CHQ-28 scoring method, based on a series of 28 questions focused on overall child health, activity limitation, emotional/behavioral difficulties, mood, relationships, and family cohesion. (Child Health Questionnaire)

SECONDARY OUTCOMES:
Parent-reported child health | 24 months
  (5-pt Likert ranging from poor to excellent) (Child Health Questionnaire)
Caregiver-reported child health care utilization, well child visits | 24 months
  Well child visits in previous 12 months (National Survey of Children's Health)
Caregiver-reported child health care utilization, sick clinic visits | 24 months
  Sick clinic visits in previous 12 months (National Survey of Children's Health)
Caregiver-reported child health care utilization, emergency room visits | 24 months
  Emergency room visits in previous 12 months (National Survey of Children's Health)
Caregiver-reported child health care utilization, hospitalization | 24 months
  Hospitalizations in previous 12 months (National Survey of Children's Health)
Usual source of care | 24 months
  Whether a child has a usual source of care when they are ill or when a parent/caregiver needs advice about their health (National Survey of Children's Health)
Forgone health care | 24 months
  Caregiver report of whether the child needed but did not receive medical, mental health, dental, or vision care in the previous 12 months (National Survey of Children's Health)
Difficulty paying medical bills | 24 months
  Difficulty paying medical bills in the previous 12 months (National Survey of Children's Health)
Uninsurance or gaps in insurance | 24 months
  Uninsurance or gaps in insurance in the previous 12 months (National Survey of Children's Health)
Average sleep duration | 24 months
  Average sleep duration in the previous week (National Survey of Children's Health)
Time spent playing outdoors, weekdays | 24 months
  Time spent playing outdoors on weekdays (National Survey of Children's Health)
Time spent playing outdoors, weekends | 24 months
  Time spent playing outdoors on weekends (National Survey of Children's Health)
Screen time | 24 months
  Screen time (National Survey of Children's Health)
Perceived neighborhood cohesion | 24 months
  Perceived neighborhood cohesion (National Survey of Children's Health)
Perceived safety of child in neighborhood | 24 months
  Perceived safety of child in neighborhood (National Survey of Children's Health)
Parenting: Difficulty caring for child | 24 months
  Parenting: Difficulty caring for child (National Survey of Children's Health)
Parenting: Child bothers parent | 24 months
  Parenting: Child bothers parent (National Survey of Children's Health)
Parenting: Anger with child | 24 months
  Parenting: Anger with child (National Survey of Children's Health)
Parenting: Handling the day-to-day demands of raising children | 24 months
  Parenting: Handling the day-to-day demands of raising children (National Survey of Children's Health)
School attendance | 24 months
  School attendance, based on Philadelphia school district data (Proportion of school days attended, internally developed)
School performance | 24 months
  School performance, based on Philadelphia school district data (Grade point average over previous 12 months, internally developed)
Rate of preterm birth | 24 months
  Rate of preterm birth (birth < 37 weeks of gestation age), based on Pennsylvania birth certificate data
Rate of low birthweight | 24 months
  Rate of low birthweight (birthweight <2000 grams), based on Pennsylvania birth certificate data
Health care utilization: emergency room visits | 24 months
  Health care utilization: emergency room visits in the previous we months, based on Children's Hospital of Philadelphia EHR data
Health care utilization: hospitalizations | 24 months
  Health care utilization: hospitalizations in the previous 12 months, based on Children's Hospital of Philadelphia EHR data

CONTACTS AND LOCATIONS:
Overall Officials: Atheendar Venkataramani, MD, PhD, Principal Investigator — University of Pennsylvania; Eugenia South, MD, MSHP, Principal Investigator — University of Pennsylvania; Aditi Vasan, MD, MSHP, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT05760001/Prot_SAP_001.pdf